CLINICAL TRIAL: NCT06429150
Title: Frontline Management of High-Risk Multiple Myeloma or Plasmacytoma With BCMA and GPRC5D Combination CAR-T Cell Therapy
Brief Title: Frontline Combination CAR-T Cell Therapy for Multiple Myeloma or Plasmacytoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Collaborators: The No.2 Clinical Hospital of the Ministry of Health (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-24001
Record Dates: First submitted 2024-05-14; First posted 2024-05-24 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Multiple Myeloma; Plasmacytoma
Keywords: multiple myeloma; chimeric antigen receptor; BCMA; GPRC5D
MeSH Terms: conditions — Multiple Myeloma; Plasmacytoma | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T cells to treat MM (Experimental)
  Interventions: Biological: CAR-T cells

INTERVENTIONS:
Biological: CAR-T cells — Infusion of multi-CAR-T cells

SUMMARY:
The aim of this clinical trial is to assess the feasibility, safety, and efficacy of CAR-T cell therapy targeting multiple cancer cell antigens in high-risk multiple myeloma or plasmacytoma as part of a frontline treatment regimen for patients. Another goal of the study is to learn more about the persistence and function of these CAR-T cells in the body.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is the second most common malignant hematological cancer in the world, which begins with the malignant proliferation of plasma cells in bone marrow. It has been a difficult disease to treat, and most patients will eventually relapse, especially for those with high-risk genotypes. At present, the therapeutic drugs for MM include glucocorticoids, cytotoxic drugs, immunosuppressants, protease inhibitors, monoclonal antibodies and cell therapies. Among those, immunotherapy has been proven to be a revolutionary treatment with great potential of curing this disease. The frequently targeted MM antigens include CD38, CD138, CD19 and BCMA, and recently, GPRC5D.

BCMA, the B cell maturation antigen, also known as CD269 or TNFRSF17, is a member of tumor necrosis factor receptor superfamily, which is highly expressed on the surface of plasma cells and partially expressed on plasma cell-like dendritic cells. It has been an ideal target for MM immunotherapy.

GPRC5D, the G-protein-coupled receptor C57 subtype D and a seven-transmembrane protein, is highly expressed on the surface of plasma cells but not in other healthy cells, and thus it has become a potential target for the treatment of MM. The expression of GPRC5D is unrelated to BCMA, so the combination therapy targeting these antigens may bring a complementary and synergistic therapeutic outcome in patients.

This trial is aimed to test the safety and efficacy of combining these different CAR-T cells targeting BCMA and GPRC5D, and in combination with well-established therapeutics as a frontline treatment for the high-risk MM or plasmacytoma patients. Another goal of this study is to investigate the persistence and function of these CAR-T cells in the body.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with multiple myeloma or plasmacytoma
* Strictly complete remission (sCR) is a treatment goal
* Expected survival > 12 weeks
* After prior auto-SCT is eligible regardless of other prior therapies
* Adequate venous access for apheresis, and no other contraindications for leukapheresis
* Voluntary informed consent is given and commitment to continued follow-up

Exclusion Criteria:

* Pregnant or lactating women
* Uncontrolled active infection
* Active HIV, hepatitis B or hepatitis C infection
* Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary.
* Any medical conditions that may preclude participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-11 (Actual); Primary Completion 2027-07-11 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with treatment related adverse effects | 1 month
  The percentage of participants with treatment-related adverse events, as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Anti-tumor activity of the fourth generation multiple CAR-T cells after infusion | 1 year
  Anti-tumor activity of the fourth generation multiple CAR-T cells after infusion by measuring the CAR copies in the blood
Anti-tumor activity of fourth generation multiple CAR-T cells in patients with high-risk MM or plasmacytoma | 1 year
  Anti-tumor activity of fourth generation multiple CAR-T cells in patients with high-risk MM or plasmacytoma by examination of known tumor indicators

CONTACTS AND LOCATIONS:
Locations (2):
- Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong, China
- Hematologist of the Regional Hematology Center in Clinical Hospital No. 2 of the Ministry of Health, Vladivostok, Russia

IPD SHARING:
Plan to Share IPD: No